CLINICAL TRIAL: NCT01300702
Title: Identification of Neuropathic Pain in the Acute Post Operative Phase Following Thoracotomy
Brief Title: Neuropathic in the Acute Post Operative Phase
Status: Terminated | Type: Observational
Why Stopped: recruitment problems
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Section for Surgical Pathophysiology (Ambiguous); Section of Acute Pain Management and Palliative Medicine (Unknown); Multidisciplinary Pain Centre (Unknown); Innovative Medicines Initiative (Other)
Responsible Party: MD, Kim Wildgaard, Section for Surgical Pathophysiology 4074
Other Study IDs: H4-2010-118#1
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lung cancer surgery: Patients undergoing thoracotomy for lung cancer

SUMMARY:
Investigation of thermal thresholds and sensory mapping to thermal stimuli

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old

Exclusion Criteria:

* do not under stand Danish
* cognitive reduction
* previous thoracic surgery
* Pregnant or nursing
* inability to cooperate to pain scoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients undergoing thoracotomy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pain | 14 days
  pain intensity
quantitative sensory testing (QST) | 14 days
  thermal thresholds assesses via QST
Neuropathic pain | 14 days
  is the pain considered neuropathic

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, MD, Study Chair — Section for Surgical Pathophysiology; Kim Wildgaard, MD, Principal Investigator — Section for Surgical Pathophysiology
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Section for Surgical Pathophysiology 4074, Copenhagen